CLINICAL TRIAL: NCT00103012
Title: The Influence of Concurrent Administration of Echinacea Purpurea, Ginkgo Biloba, or Panax Ginseng on the Steady State Pharmacokinetic Profile of Lopinavir/Ritonavir in Healthy Volunteers
Brief Title: Drug Interactions of Echinacea, Ginseng, and Ginkgo Biloba Taken With Lopinavir/Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 050082; 05-CC-0082
Record Dates: First submitted 2005-02-05; First posted 2005-02-07 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Antiretrovirals; Protease Inhibitors; Herbal Supplements; Drug Interactions; Metabolism; Healthy Volunteer; HV
MeSH Terms: interventions — Ginkgo Extract; Echinacea extract; Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Effect of G. Biloba on LPV disposition (Experimental): The primary outcome measurement for each study arm is the change in lopinavir area under the concentration versus time curve (AUC) after two weeks administration of an herbal preparation (Ginkgo Biloba).
  Interventions: Drug: Gingko Biloba
- Effect of Echinacea on LPV disposition (Experimental): The primary outcome measurement for each study arm is the change in lopinavir area under the concentration versus time curve (AUC) after two weeks administration of an herbal preparation (Echinacea purpurea).
  Interventions: Drug: Echinacea purpurea
- Effect of P. ginseng on LPV disposition (Experimental): The primary outcome measurement for each study arm is the change in lopinavir area under the concentration versus time curve (AUC) after two weeks administration of an herbal preparation (Panax ginseng).
  Interventions: Drug: Panax ginseng

INTERVENTIONS:
Drug: Gingko Biloba — Ginkgo Biloba 120 mg twice daily for 14 days
  Arms: Effect of G. Biloba on LPV disposition
Drug: Echinacea purpurea — Echinacea purpurea 500 mg three times daily for 14 days
  Arms: Effect of Echinacea on LPV disposition
Drug: Panax ginseng — Panax ginseng 500 mg twice daily
  Arms: Effect of P. ginseng on LPV disposition

SUMMARY:
This study will examine the interaction of the HIV combination medication lopinavir/ritonavir with the herbal products echinacea, ginseng, and ginkgo biloba. Patients with HIV infection often take herbal products and dietary supplements in addition to their doctor-prescribed medicines to treat the disease, lessen the side effects of anti-viral drugs, and improve their overall well being. Alternative medicines such as these may, however, interfere with the elimination of lopinavir/ritonavir from the body, causing either higher or lower blood levels of these drugs than would be expected. This study will assess in healthy subjects any potential harms of taking echinacea, ginseng, or ginkgo biloba together with lopinavir/ritonavir.

Healthy normal volunteers between 18 and 50 years of age may be eligible for this study. Candidates are screened with a history, physical examination, and blood tests, including an HIV test and a pregnancy test for women. Pregnant women are excluded from the study. Participants come to the NIH Clinical Center after fasting overnight for the following procedures:

Visits 1 and 2: A catheter (plastic tube) is placed in an arm vein to collect blood samples. After the first sample is drawn, the subject takes 8 mg of midazolam syrup and two fexofenadine tablets. Midazolam is a sedative, and fexofenadine (Allegra) is a medicine used to treat allergies. Subjects are given breakfast an hour after taking the drugs. Blood samples are collected at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8 and 24 hours after taking the drugs to measure blood levels of fexofenadine. An extra sample is collected at the 4-hour mark to measure the midazolam level. The catheter is removed after the 8-hour blood draw and subjects are dismissed home. They return the following morning (visit 2) for the 24-hour blood draw.

Visit 3: From 7 to 28 days after visit 1, subjects begin taking lopinavir/ritonavir capsules twice a day by mouth for a total of 29.5 days. On day 15 they return to the clinic for lopinavir/ritonavir blood levels as were done for fexofenadine, except that samples are collected once before breakfast and then at 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after the lopinavir/ritonavir dose. An extra sample is collected for routine tests. The catheter is removed after the 12-hour draw and the subject is dismissed home.

The next morning, subjects begin taking one of the following: echinacea 500 mg 3 times a day; ginkgo biloba 120 mg twice a day; or ginseng 500 mg 3 times a day for 28 days.

Visit 4: On the last day of taking lopinavir/ritonavir, subjects return to the clinic again for blood level measurements of these drugs as on visit 3, except that the catheter is removed and the subject dismissed home after the 8-hour blood draw.

Visits 5 and 6: On the last day of taking the herbal supplement, subjects return to the clinic for repeat measurement of fexofenadine and midazolam levels, as described in visits 1 and 2. At the final visit (visit 6) an additional blood sample is collected for repeat laboratory testing.

...

DETAILED DESCRIPTION:
Patients with HIV commonly use herbal products and dietary supplements in addition to medications prescribed by their physicians. Up to 73% of patients with HIV have reported using some form of complementary or alternative medicine. As such, the potential for clinically significant drug interactions between herbs and antiretrovirals is becoming increasingly appreciated. Despite this awareness, little is known about the effect of commonly used herbal products, such as echinacea, ginkgo biloba, and ginseng, on antiretroviral pharmacokinetics. Interacting herbal supplements have the potential to alter protease inhibitor (PI) plasma concentrations, as has been shown with St. John's Wort and garlic. Drug interactions may potentially increase antiretroviral concentrations, putting patients at risk for toxicities, or lower drug concentrations below the threshold of viral susceptibility, putting patients in jeopardy of antiretroviral failure. The protease inhibitors lopinavir and ritonavir both rely principally on cytochrome P450 (CYP) 3A4 metabolism for their elimination. In addition, both drugs are substrates for the transport protein p-glycoprotein (P-gp), which may also contribute to their distribution and elimination.

The primary purpose of this investigation is to determine whether the herbal supplements Echinacea purpurea, ginkgo biloba, and Panax ginseng alter the pharmacokinetic properties of the HIV protease inhibitor (PI) lopinavir, administered as the PI combination lopinavir/ritonavir (LPV/r). This is an open label pharmacokinetic study that will be performed on an outpatient basis. A total of 42 study participants who have met inclusion criteria will be sequentially divided into one of 3 groups, such that 14 subjects each will receive LPV/r alone and in combination with either E. purpurea, G. biloba, or P. ginseng.

Subjects will begin taking LPV/r (400mg/100mg twice daily x 29.5 days), returning to the NIH on Day 15 of dosing for post-dose plasma collection and determination of lopinavir and ritonavir concentrations. On Day 16 participants will begin taking either E. purpurea (500mg, three times daily), G. biloba extract (120 mg, twice daily), or P. ginseng (500 mg, twice daily) for 28 days. On the 30th day of LPV/r (Day 15 of the herb), subjects will return to the NIH where they will take their final LPV/r dose and then have their plasma collected for determination of lopinavir concentrations. Data from this investigation will determine whether echinacea, ginseng, or ginkgo biloba supplements alter the pharmacokinetics of lopinavir.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females between the ages of 18 and 50 years.
  2. Healthy by medical history and physical exam.
  3. Laboratory values within established guidelines for participation in clinical studies: AST less than or equal to 2 times the ULN; SCr less than or equal to ULN; hemoglobin equal to or greater than 11 g/dL (for both males and females).
  4. Ability to abstain from ingesting fruit juice during pharmacokinetic sampling periods (a total of 2 study days), and abstain from eating grapefruit or drinking grapefruit juice during the entire study period.
  5. Negative serum or urine pregnancy test for females of child-bearing potential.
  6. Females of child-bearing potential who are able and willing to practice abstinence or use non-hormonal effective methods of birth control during the study, such as condoms or diaphragms.

EXCLUSION CRITERIA:

1. Concomitant routine therapy with any prescription, over-the-counter, herbal, or holistic medications, including oral contraceptives, for 30 days prior to study participation. Intermittent use of any medication within 30 days prior to screening will be considered case by case by the principal investigator and the medically accountable investigator.

   * Concomitant therapy (chronic or intermittent) with any prescription, over-the-counter, or herbal drugs (including tinctures, foods, beverages, and gum) will not be allowed during the study duration, including any intermittent use of allergy medication.
   * Intermittent use of acetaminophen, non-steroidal anti-inflammatory medications (i.e. ibuprofen), and loperamide will be allowed during the study, but should not be taken on the days of pharmacokinetic blood sampling.
   * A daily multivitamin with minerals will be allowed during the study.
2. Inability to obtain venous access for blood sample collection.
3. The presence or history of any of the following: diabetes mellitus (clinical diagnosis based on current guidelines, HIV infection, active tuberculosis, cardiac disease (eg. Hypertension [SBP greater than 140 mmHG or DBP greater than 90 mmHG], heart failure, arrhythmia, etc.), renal disease, hepatitis or hepatic impairment, pancreatitis, bleeding disorders, internal bleeding (such as gastrointestinal or intracranial), respiratory disease (eg. asthma requiring maintenance pharmacologic therapy, chronic obstructive pulmonary disease, etc.), peptic ulcer disease, osteoporosis, osteonecrosis, atopy or atopic dermatitis, hormone sensitive cancers or conditions, organ transplant, seizure disorders, schizophrenia or other psychiatric illnesses that may interfere with the subject's ability to participate in the study, or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators.
4. Plans for elective surgery during the investigation or within 1 month following completion for subjects in the gingko biloba arm of the study.
5. Positive serum or urine pregnancy test or breastfeeding female.
6. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
7. Drug or alcohol abuse that may impair safety or adherence (more than 3 alcoholic drinks per day, on a daily basis).
8. History of intolerance or allergic reaction to any products containing echinacea, ginkgo biloba extract, or ginseng (including pills, tinctures, foods, beverages, and gum).
9. History of intolerance or allergic reaction to lopinavir, ritonavir, midazolam, or fexofenadine.
10. History of atopy including atopic dermatitis, bronchial asthma, multiple food allergies, or severe recurring allergic rhinitis.
11. Fasting total cholesterol greater than 240 mg/dL or fasting triglycerides greater than 400 mg/dL.
12. Use of nicotine-containing tobacco products, including cigarettes and chewing tobacco.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2005-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Penzak, Pharm.D., Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fairfield KM, Eisenberg DM, Davis RB, Libman H, Phillips RS. Patterns of use, expenditures, and perceived efficacy of complementary and alternative therapies in HIV-infected patients. Arch Intern Med. 1998 Nov 9;158(20):2257-64. doi: 10.1001/archinte.158.20.2257. PMID 9818806
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257
- [Background] Risa KJ, Nepon L, Justis JC, Panwalker A, Berman SM, Cinti S, Wagener MM, Singh N. Alternative therapy use in HIV-infected patients receiving highly active antiretroviral therapy. Int J STD AIDS. 2002 Oct;13(10):706-13. doi: 10.1258/095646202760326471. PMID 12396542
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-CC-0082.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy human volunteers were recruited to participate in this study throughout the course of the investigation (2005-2010).
Groups:
- Influence of Ginkgo Biloba on Lopinavir/Ritonavir Disposition: Lopinavir + ritonavir (x 2 weeks), midazolam (single dose), and fexofenadine (single dose) pharmacokinetics determined before, and after 14-28 days of Ginkgo Biloba administration (120 mg two times daily) to healthy human volunteers.
- Influence of Echinacea on Lopinavir/Ritonavir Disposition: Lopinavir + ritonavir (x 2 weeks), midazolam (single dose), and fexofenadine (single dose) pharmacokinetics determined before, and after 14-28 days of Echinacea(500 mg three times daily).
- Influence of Panax Ginseng on Lopinavir/Ritonavir Disposition: Lopinavir (x 2 weeks), midazolam (single dose), and fexofenadine (single dose) pharmacokinetics determined before, and after 14-28 days of Panax ginseng (500 mg twice daily).
Period: Overall Study
Arm/Group | Influence of Ginkgo Biloba on Lopinavir/Ritonavir Disposition | Influence of Echinacea on Lopinavir/Ritonavir Disposition | Influence of Panax Ginseng on Lopinavir/Ritonavir Disposition
Started | 17 | 14 | 16
Completed | 14 | 13 | 12
Not Completed | 3 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Subject non-compliant with medications | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influence of Ginkgo Biloba on Lopinavir/Ritonavir Disposition | Influence of Echinacea on Lopinavir/Ritonavir Disposition | Influence of Panax Ginseng on Lopinavir/Ritonavir Disposition | Total
Number analyzed (Participants) | 17 | 14 | 16 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 16 | 47
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (9.3) | 33 (8.5) | 32 (6.4) | 33 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 4 | 18
  Male | 8 | 9 | 12 | 29
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Lopinavir Pharmacokinetics When Administered Alone and in Combination With Three Different Herbal Supplements: Ginkgo Biloba, Panax Ginsing, and Echinacea Purpurea.
Description: The outcome measurement for each study arm is the change in lopinavir area under the concentration versus time curve (AUC) after two weeks administration of an herbal preparation (Ginkgo Biloba, Echinacea purpurea, or Panax Ginseng).
Time Frame: 2 weeks
Population: Data was analyzed from all subjects who completed a particular sampling period.
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*hr/mL
Groups:
- Influence of Ginkgo Biloba on Lopinavir Disposition: Lopinavir pharmacokinetics (administered as lopinavir-ritonavir X 2 weeks) determined before, and after 14 days of Ginkgo Biloba administration (120 mg two times daily) to healthy human volunteers.
- Influence of Echinacea on Lopinavir Disposition: Lopinavir (administered as lopinavir-ritonavir X 2 weeks)pharmacokinetics determined before, and after 14 days of Echinacea purpurea administration (500 mg three times daily) to healthy human volunteers.
- Influence of Panax Ginseng on Lopinavir Disposition: Lopinavir (administered as lopinavir-ritonavir X 2 weeks)pharmacokinetics determined before, and after 14-28 days of Panax ginseng (500 mg twice daily).
Arm/Group | Influence of Ginkgo Biloba on Lopinavir Disposition | Influence of Echinacea on Lopinavir Disposition | Influence of Panax Ginseng on Lopinavir Disposition
Number analyzed (Participants) | 14 | 13 | 12
mcg*hr/mL | 1.02 [0.67 to 1.38] | 0.96 [0.83 to 1.10] | 1 [0.3 to 2]

ADVERSE EVENTS:
Arm/Group | Influence of Ginkgo Biloba on Lopinavir/Ritonavir Disposition | Influence of Echinacea on Lopinavir/Ritonavir Disposition | Influence of Panax Ginseng on Lopinavir/Ritonavir Disposition
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 2/17 | 13/14 | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influence of Ginkgo Biloba on Lopinavir/Ritonavir Disposition (N=17) | Influence of Echinacea on Lopinavir/Ritonavir Disposition (N=14) | Influence of Panax Ginseng on Lopinavir/Ritonavir Disposition (N=16)
diarrhea (Gastrointestinal disorders) | 1 (2) | 11 (26) | 9 (22)
dysmenorrhea (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1)
electrolyte imbalance (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3)
headache (Nervous system disorders) | 0 (0) | 2 (2) | 7 (10)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (7) | 2 (5)
acute sore throat (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
sinus congestion (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
decreased concentration (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
taste alterations (General disorders) | 0 (0) | 1 (1) | 0 (0)
anorexia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
cough (General disorders) | 0 (0) | 1 (1) | 0 (0)
fever (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
generalized pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
common cold (General disorders) | 1 (2) | 0 (0) | 1 (1)
decreased serum albumin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
decreased absolute neutrophil count (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
elevated ALT (SGPT) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
elevated AST (SGOT) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
elevated serum bilirubin (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3)
fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3)
dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
decreased hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes